CLINICAL TRIAL: NCT01909479
Title: A Phase 3, Multicenter Study Designed To Evaluate The Efficacy And Safety Of A Long Acting hGH Product (MOD-4023) In Adult Subjects With Growth Hormone Deficiency
Brief Title: A Phase 3, Multicenter Study To Evaluate The Efficacy And Safety Of MOD-4023 In Adults With Growth Hormone Deficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Main Study was completed. LT-OLE was discontinued as sufficient safety data has been generated.
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-4-005; 2013-000830-37 (EudraCT Number)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — MOD-4023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOD-4023 (Experimental)
  Interventions: Drug: MOD-4023
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MOD-4023 — Individualized once weekly dose of MOD-4023
  Arms: MOD-4023
Other: Placebo — Once weekly administration of placebo
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, parallel-group, multicenter study in adult subjects with GHD to assess the safety and efficacy of a long-acting, once weekly injection of modified hGH (MOD-4023).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the age of 23 to 70 years old at screening, inclusive
* GHD subjects as defined in the Consensus guidelines for the diagnosis and treatment of adults with GH deficiency II (2007).
* No r-hGH replacement therapy or use of GH secretagogues for at least 9 months with any registered or investigational r-hGH or GH secretagogue product.
* The IGF-I level at screening ≤-1 SDS of the age and sex normal ranges according to the central laboratory measurements
* Subjects who are on a stable diet and exercise regime and do not have plans to modify their diet or exercise for at least 12 months
* Subject had a DXA screening and the results are interpretable according to the study plan.

Exclusion Criteria:

* Women who are pregnant or breast-feeding (at least 6 months delay from childbirth or lactation)
* Evidence of growth benign intracranial tumor within the last 12 months (determined by comparing a previous MRI to a new one obtained no more than 6 months prior to study entry to clarify dynamics of growth).
* History of any cancer. Exceptions to this exclusion criterion include resected in situ carcinoma of the cervix and squamous cell or basal cell carcinoma of the skin with complete local excision. Patients with GHD attributed to treatment of intracranial malignant lesions in childhood or adulthood (or, tumors) or leukemia may also be enrolled into the study provided that a recurrence-free survival period of at least 5 years is well documented in the study record.
* Signs of intracranial hypertension at screening
* Heart insufficiency, NYHA class > 2 (Appendix B)
* History of overt diabetes mellitus (including currently treated, well-controlled DM) defined according to the American Diabetes Association (ADA) Criteriaa. A history of gestational diabetes, resolved after childbirth, is not exclusionary.
* History of Acromegaly

Ages: 23 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-06; Primary Completion 2016-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Opko Biologics, Kiryat Gat, Israel

RESULTS

PARTICIPANT FLOW:
Period: From Baseline to Week 26
Arm/Group | MOD-4023 | Placebo
Started | 135 | 67
Completed | 129 | 58
Not Completed | 6 | 9
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Site and study closed by PI | 0 | 1
Period: 26 - 52 Weeks
Arm/Group | MOD-4023 | Placebo
Started (One patient withdrew consent after completing Period 1) | 128 | 58
Completed | 125 | 56
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: 52 Weeks to End of Study
Arm/Group | MOD-4023 | Placebo
Started | 111 (Not all of the participants that completed the previous period continued on in the study) | 50 (Not all of the participants that completed the previous period continued on in the study)
Completed | 83 | 35
Not Completed | 28 | 15
Not completed — Withdrawal by Subject | 18 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive disease | 1 | 1
Not completed — Personal reasons | 2 | 1
Not completed — Sponsor's decision | 1 | 1
Not completed — Study termination by sponsor | 0 | 1
Not completed — Lack of contact | 1 | 0
Not completed — Occurrence of malignancy | 1 | 0
Not completed — Diabetes not controlled | 0 | 1

BASELINE CHARACTERISTICS:
Population: 202 subjects met the study's eligibility criteria and were randomized to either MOD-4023 or placebo. Only 198 subjects actually treated and included in the efficacy analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | MOD-4023 | Placebo | Total
Number analyzed (Participants) | 133 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: Year] | 43.9 (12.6) | 43.1 (12.9) | 43.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 25 | 82
  Male | 76 | 40 | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 110 | 53 | 163
  Black or African American | 1 | 2 | 3
  Asian | 15 | 8 | 23
  Other | 2 | 0 | 2
  Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 31 | 15 | 46
  Europe | 88 | 43 | 131
  East Asia | 14 | 7 | 21
Weight [Mean (Standard Deviation); unit: Kilogram] | 75.2 (15.0) | 77.8 (17.9) | 75.2 (15.0)
BMI [Mean (Standard Deviation); unit: Kilogram/meter^2] | 27.0 (3.2) | 27.7 (3.5) | 27.0 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Trunk Fat Mass, Expressed in Kilograms Measured With Dual-energy X-ray Absorptiometry, From Baseline to Week 26
Time Frame: Baseline to 26 weeks
Population: 198 of the 202 randomized subjects received treatment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 126 | 56
kg | -0.3 (1.2) | 0.1 (1.6)

2. Secondary Outcome: Change in Total Fat Mass, Expressed in Kilograms, Measured With Dual-energy X-ray Absorptiometry, From Baseline to Week 26
Time Frame: Baseline to 26 weeks
Population: 3 subjects discontinued MOD-4023 due to consent withdrawn or lost to follow-up. 2 subjects discontinued placebo due to consent withdrawn or adverse event.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 126 | 56
kg | -0.18 (2.21) | 0.00 (2.64)

3. Secondary Outcome: Change in Lean Body Mass, Expressed in Kilograms Measured With Dual-energy X-ray Absorptiometry, From Baseline to Week 26
Time Frame: Baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 126 | 56
kg | 1.3 (2.4) | 0.0 (1.6)

4. Secondary Outcome: Change in Trunk Fat Mass, Expressed in Kilograms Measured With Dual-energy X-ray Absorptiometry, From Baseline to 52 Weeks
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 125 | 55
kg | -0.2 (1.6) | -0.3 (2.1)

5. Secondary Outcome: Change in Trunk Fat Mass, Expressed as % Change From Baseline, Measured With Dual-energy X-ray Absorptiometry, From Baseline to 26 and 52 Weeks
Time Frame: 26 weeks to 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 125 | 56
percentage of change from baseline
  % Change from baseline in week 26 | -2.4 (8.5) | 0.8 (10.0)
  % Change from baseline in week 52: number analyzed (Participants) | 125 | 55
  % Change from baseline in week 52 | -1.6 (3.1) | -1.2 (2.8)

6. Secondary Outcome: Trunk Fat Mass as Percentage of Total Fat Mass From Baseline to Week 26
Time Frame: Baseline to 26 weeks
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 126 | 56
percentage of change from baseline | -1.8 (3.0) | 0.6 (2.7)

7. Secondary Outcome: Change in Biochemical Marker IGF-1
Time Frame: Baseline to 26 weeks
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | MOD-4023 | Placebo
Number analyzed (Participants) | 131 | 59
ug/L | 134.1 (42.4) | 54.5 (29.2)

ADVERSE EVENTS:
Time Frame: These events were collected throughout the duration of the study and cumulative to weeks Period 1, Baseline to 26 weeks Period 2, 26 - 52 weeks Period 3, >52 weeks to end of study **up to 2 years**
Description: AEs collected and reported for each period of the study. Period 1, Baseline to 26 weeks Period 2, 26 - 52 weeks Period 3, >52 weeks to end of study
Groups:
- MOD-4023 Period 1: MOD-4023: Individualized once weekly dose of MOD-4023 (Period 1)
- Placebo Period 1: Placebo: Once weekly administration of placebo (Period 1. Only till week 26). Open label once weekly dose of MOD-4023 thereafter
- MOD-4023 Period 2 (Treatment Assignments at Period 1): MOD-4023: Individualized once weekly dose of MOD-4023 (Period 2)
- Placebo Period 2 (Treatment Assignments at Period 1); Placebo Period 3 (Treatment Assignments at Period 1): Placebo assigned and treated in Period 1. Open-label MOD-4023 treatment in Periods 2 and 3
- MOD-4023 Period 3 (Treatment Assignments at Period 1): MOD-4023: Individualized once weekly dose of MOD-4023 (Period 3).
  Period 3 was a long-term open label extension
Arm/Group | MOD-4023 Period 1 | Placebo Period 1 | MOD-4023 Period 2 (Treatment Assignments at Period 1) | Placebo Period 2 (Treatment Assignments at Period 1) | MOD-4023 Period 3 (Treatment Assignments at Period 1) | Placebo Period 3 (Treatment Assignments at Period 1)
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/65 | 0/133 | 0/65 | 0/111 | 1/50
Serious Adverse Events (participants affected / at risk) | 4/133 | 5/65 | 5/133 | 3/65 | 10/111 | 8/50
Other Adverse Events (participants affected / at risk) | 36/133 | 27/65 | 28/133 | 16/65 | 46/111 | 30/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 Period 1 (N=133) | Placebo Period 1 (N=65) | MOD-4023 Period 2 (Treatment Assignments at Period 1) (N=133) | Placebo Period 2 (Treatment Assignments at Period 1) (N=65) | MOD-4023 Period 3 (Treatment Assignments at Period 1) (N=111) | Placebo Period 3 (Treatment Assignments at Period 1) (N=50)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pituitary-dependent Cushing's syndrom (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hemianopia heteronymous (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device loosening (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 Period 1 (N=133) | Placebo Period 1 (N=65) | MOD-4023 Period 2 (Treatment Assignments at Period 1) (N=133) | Placebo Period 2 (Treatment Assignments at Period 1) (N=65) | MOD-4023 Period 3 (Treatment Assignments at Period 1) (N=111) | Placebo Period 3 (Treatment Assignments at Period 1) (N=50)
Injection site pain (General disorders) | 12 | 9 | 4 | 4 | 4 | 4
Nasopharyngitis (Infections and infestations) | 5 | 5 | 10 | 4 | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 0 | 0 | 10 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 5 | 11 | 2 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 6 | 3 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 5
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 7 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less